CLINICAL TRIAL: NCT04716075
Title: Acalabrutinib in CLL and MCL Patients Subjected to Allogeneic Hematopoietic Stem Cell Transplantation (alloSCT)
Acronym: ACALLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Polish Lymphoma Research Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLRG12
Record Dates: First submitted 2020-12-17; First posted 2021-01-20 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Chronic Lymphocytic Leukemia; Chronic Graft-versus-host-disease; Mantle Cell Lymphoma; Adverse Event; Response Rate
Keywords: acalabrutinib; Chronic Lymphocytic Leukaemia; allogeneic haematopetic cell transplantation; Chronic Graft-versus-host-disease; Minimal Residual Disease; reduced intensity conditioning; Mantle Cell Disease
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Bronchiolitis Obliterans Syndrome; Lymphoma, Mantle-Cell; Leukemia, B-Cell; Neoplasm, Residual

STUDY DESIGN:
Intervention Model Description: Multicentre, national
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acalabrutinib 2x100mg oral capsule +alloSCT (Experimental): Acalabrutinib administered 2x100mg p.o. daily for 3-6 months before alloSCT +acalabrutinib administered 2x100mg p.o. daily for 9 months after alloSCT
  Interventions: Drug: Acalabrutinib 2x100 MG Oral Capsule + alloSCT

INTERVENTIONS:
Drug: Acalabrutinib 2x100 MG Oral Capsule + alloSCT — Acalabrutinib 100 mg caps will be administered twice daily for 3-6 months before the intended alloSCT. After restarting acalabrutinib (2x100 mg daily) after the transplant procedure it will be administered for further 9 months. In patients who do not have an acceptable donor acalabrutinib will be administered until disease progression or unacceptable toxicity.

SUMMARY:
In this phase II multicenter trial we plan to use acalabrutinib before and after allogeneic hematopoietic stem cell transplantation (alloSCT) with reduced intensity conditioning (RIC) in patients with refractory/relapsed MCL and CLL with poor prognostic factors. Acalabrutinib will be used before alloSCT with the intention to reduce tumor burden and after transplant to augment disease control.

DETAILED DESCRIPTION:
In this phase II multicenter trial we plan to use acalabrutinib before and after allogeneic hematopoietic stem cell transplantation (alloSCT) with reduced intensity conditioning (RIC) in patients with refractory/relapsed MCL and CLL with poor prognostic factors. Acalabrutinib will be used before alloSCT with the intention to reduce tumor burden and after transplant to augment disease control. Since chronic GvHD is mediated by activated B lymphocytes, we also speculate that the drug as a BTK inhibitor may reduce the severity and incidence of chronic graft-versus-host disease (GvHD) after alloSCT, as it was shown for ibrutinib.

Best response to therapy and safety issues will be the primary target of this small trial (25 transplanted pts).TEAE and SAE of acalabrutinib in patients after alloSCT that was not previously assessed.

We hypothesize that this treatment will improve the efficacy of the alloSCT - this issue will be addressed by serial minimal residual disease (MRD) evaluation in peripheral blood and bone marrow. This treatment strategy could significantly improve the outcome of poor prognosis MCL and CLL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age.
2. Relapsing / refractory BTK-inhibitors naïve CLL patients meeting IWCCL criteria for requiring treatment:

   1. after 1-4 therapy lines if del 17 or p53 mutation in >10% of analyzed CLL cells (PB or BM) or
   2. after 2-4 therapy lines if high risk CLL (refractory or less than 24 months response to the last immunochemotherapy) or Confidential Page 15 of 82 Study Protocol v. 1.5 dated 06.07.2018
3. Relapsing / refractory BTK-inhibitors naïve MCL patients with measurable disease or bone marrow involvement revealed in trephine biopsy or
4. Patients fulfilling criteria 2 or 3, when ibrutinib therapy was initiated, responding to therapy
5. Patient qualified for allo SCT procedure by the transplant center participating in the trial with identified sibling donor or initiated Poltransplant search for matched unrelated donor.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Woman of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and for 2 days after the last dose of acalabrutinib and for 6 months after the transplant procedure if performed. Males who are sexually active must use highly effective methods of contraception during treatment and for 6 months after the transplant procedure if performed.
8. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
9. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information

Exclusion Criteria:

1. Patients failing 5 or more previous therapy lines
2. Prior malignancy (or any other malignancy that requires active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 5 years
3. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or Confidential Page 16 of 82 Study Protocol v. 1.5 dated 06.07.2018 any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification (NYHA). Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study.
4. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
5. Impaired hepatic function (as indicated by any of the following):

   1. Serum total bilirubin > 2.5 x upper limit of normal (ULN)
   2. Alanine amino transferase and/or aspartate amino transferase > 2.5 x ULN
   3. Alkaline phosphatase > 2.5 x ULN
6. Impaired renal function: serum creatinine > 2.5 x ULN
7. Other concurrent serious diseases that increase Hematopoietic Cell Transplantation-Comorbidity Index (HCT-CI) > 4
8. Central nervous system involvement with CLL
9. Known history of drug-specific hypersensitivity or anaphylaxis to study drug (including active product or excipient components).
10. Active bleeding, history of bleeding diathesis (eg, hemophilia or von Willebrand disease).
11. Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura).
12. Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening.
13. Requiring or receiving a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer (see appendix 3 for a complete list) Confidential Page 17 of 82 Study Protocol v. 1.5 dated 06.07.2018
14. Requiring or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon) within 7 days of first dose of study drug.
15. Requiring proton pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
16. Prothrombin time/INR or aPTT (in the absence of Lupus anticoagulant) > 2x ULN.
17. History of significant cerebrovascular disease or event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug.
18. Major surgical procedure within 30 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
19. Known history of infection with HIV or any active uncontrolled systemic infection
20. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded.

    Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded.
21. ANC < 500/μl, Platelets < 20 000/μl, and hemoglobin < 8 g/dl
22. Breastfeeding or pregnant.
23. Concurrent participation in another therapeutic clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Response Rate | through study completion on average 27 months
  Nr of patients with partial and complete response (PR and CR),
Response to therapy Minimum residual disease CR (MRD CR) rate | through study completion on average 27 months
  Nr of patients with minimum residual disease CR (MRD CR) assessed by flow cytometry in peripheral blood (PB) and bone marrow (BM)
Adverse event/serious adverse event incidence | acalabrutinib completion or discontinuation plus 30 days of the last acalabrutinib dose
  Incidence of adverse events per system

SECONDARY OUTCOMES:
Non-relapse mortality | through study completion on average 27 months
  Nr of patients who died being in continuous remission
Relapse incidence | through study completion on average 27 months
  Nr of patients with return of a disease or the signs and symptoms of a disease after a period of improvement
Progression free survival | through study completion on average 27 months
  Nr of days from assignment in a clinical trial to disease progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Giebel, Prof., Study Chair — Polish Lymphoma Research Organization
Locations (6):
- Poland (6):
  - Szpital Kliniczny Przemienienia Pańskiego, Oddział Hematologii i Transplantacji Szpiku, Poznan, Greater Poland Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Narodowy Intytut Onkologii im. M. Skłodowskiej-Curie Oddział w Krakowie, Pododdział Leczenia Nowotworów Układu Chłonnego, Krakow, Małopolska
  - Klinika Transplantacji Szpiku i Onkohematologii; Centrum Onkologii Instytut im. M.Sklodowskiej-Curie, Oddz. w Gliwicach, Gliwice, Silesian Voivodeship
  - Narodowy Instytut Onkologii - im. Marii Skłodowskiej- Curie -Państwowy Instytut Badawczy Klinika Nowotworów Układu Chłonnego, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wrocławiu Katedra i Klinika Hematologii, Nowotworów Krwi i Transplantacji Szpiku Uniwersytetu Medycznego, Wroclaw

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT04716075/Prot_SAP_000.pdf